CLINICAL TRIAL: NCT00519545
Title: Prayer as a Possible Adjuvant Treatment for Breast Cancer - A Randomized Partially Blinded Controlled Clinical Trial Evaluating the Effect of Prayer on Humoral and Biochemical Parameters in Stage I-IV Breast Cancer
Brief Title: Prayer as a Possible Adjuvant Treatment for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southwestern Regional Medical Center (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Dan Nixon, M.D., Cancer Control Center of Charleston, Charleston South Carolina
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: CTCA 05-04
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Breast Neoplasms
Keywords: breast; cancer; stage; one; four
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Faith Healing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): scripted prayer group (intervention group)
  Interventions: Behavioral: Prayer
- 2 (No Intervention): no prayer intervention group (non-intervention group)

INTERVENTIONS:
Behavioral: Prayer — Data collection on physiological biomarkers
  Arms: 1

SUMMARY:
The goal of this study is to help determine the biochemical mechanisms underlying previously demonstrated health benefits of prayer, and to track humoral changes in various prayer activities.

DETAILED DESCRIPTION:
The purpose of this pilot study is to investigate certain biological mechanisms that may underlie the beneficial effects seen among cancer patients who pray. It will evaluate the effect of prayer on humoral (including biochemical/physiological inflammatory/immune) parameters, monitor changes in cancer related biomarkers and evaluate the effect of prayer on blood pressure, quality of life, health and dietary habits in relation to prayer activities, using validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Primary histological diagnosis of Stage I-IV breast cancer.
2. Initial diagnosis of breast cancer within 5 year of study enrollment.
3. Not currently receiving chemotherapy or radiation therapy. Hormone therapy is allowed.
4. Life expectancy of at least 12 months.
5. ECOG performance status of 0, 1, or 2.
6. Willing to sign informed consent indicating that they are aware of the investigational nature of the study and the randomized study design.
7. Willing to comply with monthly follow-up phone calls.
8. Willing to complete questionnaires at regular oncology clinic visits.
9. Able to read write & understand English.

Exclusion Criteria:

1. Concurrent treatment with chemotherapy or radiation therapy
2. Less than 3 months since last dose of chemotherapy or radiation therapy.
3. Breast cancer diagnosis more than 5 years prior to study enrollment
4. Less than 21 or greater than to 80 years old.
5. Life threatening or severe concurrent non-malignant conditions.
6. Uncontrolled diabetes mellitus.
7. Severe heart disease.
8. Severe liver disease. Severe lung disease.
9. History of smoking within 5 years of study enrollment.
10. Psychological or psychiatric disorder that would interfere with study compliance.
11. History of missed appointments or poor medical compliance.
12. Inability to understand instructions on how to complete a questionnaire.
13. No access to a phone.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
A. Evaluate the effect of prayer on humoral (including biochemical/physiological inflammatory/immune) parameters approximately every three months at the subjects routine oncology visit. | 2 years
B. Monitor changes in cancer- related biomarkers, and evaluate these changes in relation to the participants' prayer activities as recorded since the previous oncology visit. | 2 years
C. Evaluate the effect of prayer on blood pressure, quality of life, health and dietary habits in relation to prayer activities, using validated questionnaires. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ray, MD, Principal Investigator — Cancer Treatment Centers of America; Petra Ketterl, MD, Principal Investigator — Cancer Treatment Centers of America at Southwestern Regional Medical Center; Percy McCray, Rev., Principal Investigator — Cancer Treatment Centers of America; Michael Langham, Rev., Principal Investigator — Cancer Treatment Centers of America at Southwestern Regional Medical Center; Daniel Nixon, MD, Principal Investigator — Cancer Control Center of Charleston
Locations (1):
- Cancer Treatment Centers of America at Southwestern Regional medical Center, Tulsa, Oklahoma, United States